CLINICAL TRIAL: NCT05174104
Title: Impact of Vestibular Rehabilitation on Metabolic Aspects and Chronobiological Behavior
Brief Title: Metabolic and Chronobiological Changes in Vestibular Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uniter Onlus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UniterVestib
Record Dates: First submitted 2021-12-10; First posted 2021-12-30 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2021-12

CONDITIONS: Vestibular Disorder; Metabolic Disease; Sleep Disorder
MeSH Terms: conditions — Vestibular Diseases; Metabolic Diseases; Sleep Wake Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Vestibular Rehabilitation (Experimental): This group will undergo a 4 weeks of vestibular rehabilitation in the first month and then it will be only followed up in the second month
  Interventions: Procedure: Vestibular Rehabilitation
- Delayed Vestibular Rehabilitation (Experimental): This group will be followed-up for the first month and the it will undergo 4 weeks of vestibular rehabilitation in the second month
  Interventions: Procedure: Vestibular Rehabilitation

INTERVENTIONS:
Procedure: Vestibular Rehabilitation — The home exercise schedule consists of a patient-tailored association of adaptation (without and with the target moving on pitch and yaw planes for 1 min each three times per day), substitution, habituation, and balance and gait exercises. All the unilateral vestibular hypofunction patients will be followed in the clinic twice a week for 4 weeks for 30-45 min and evaluated for adherence. Between supervised sessions, patients will perform a twice-daily home exercise plan for a total of 30-40 min/day

SUMMARY:
The aim of the present study is to evaluate the impact of vestibular rehabilitation on metabolic aspects when evaluated by means of bioelectrical impedenzometry analysis, smart watch device and actigraphy in a group of vestibular hypofunction patients previously studied by means of video head impulse test, posturography and clinical validated scales

DETAILED DESCRIPTION:
Recent advances in the field of vestibular-related disorders demonstrated that such conditions may interfere on different pathways underpinning metabolic behaviour, daily life activities and also chronotype behaviour. However, no studies evaluated how vestibular rehabilitation procedures - well established in literature - may interfere on these vestibular-related disorders. On the other side, recent advances in portable bioelectrical impedenzometry devices, smart watches devised to evaluate energy expenditure during daily life activities and actigraphy devices demonstrated to be useful in continuously monitoring different aspects of metabolic, activity and sleep behaviour.

Thus, the aim of the present study is to evaluate the impact of vestibular rehabilitation on metabolic aspects when evaluated by means bioelectrical impedenzometry analysis, smart watch device and actigraphy in a group of vestibular hypofunction patients previously studied by means of video head impulse test, posturography and clinically validated scales

ELIGIBILITY:
Inclusion Criteria:

* unilateral vestibular hypofunction achieved according to accepted criteria, by bithermal caloric irrigation, showing at least 25% reduced vestibular response on one side when calculated by means of Jongkees' formula, 3 months or later after symptom onset. In order to avoid confounding factors, and following previous experiences, only subjects presenting with a concurrent reduction in vestibulo-ocular reflex (VOR) gain when studied by means of video head impulse test will be included in this study.

Exclusion Criteria:

* History of falls, cardiovascular, metabolic, rheumatologic, orthopedic, or other neurological conditions, liver or renal abnormalities.
* pregnancy or breastfeeding.
* Neurological and neuro-psychiatric diseases
* insulin-dependent diabetes, vitamin deficiencies, hypothyroidism, lung diseases, hepatitis, chronic kidney failure, and Cushing syndrome
* medication possibly impacting on cochleo-vestibular function or with a history of drug or alcohol addiction
* inability to understand and agree to the examination procedures.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Fat Mass Percentage | one month
  Fat mass percentage will be calculated by using single-frequency BIA with eight-point tactile electrodes (Omron HBF-500 BIA, Omron Medizintechnik, Mannheim, Germany), whose reliability with DXA and MRI measurements was previously demonstrated will be used. This device uses an AC of 500 µA with a single frequency of 50 kHz and eight electrodes in a tetrapolar arrangement, requiring the subject to stand on metal footpads in bare feet and grasp a pair of electrodes fxed on a handle, with arms extended in front of the chest.
Muscle Mass Percentage | one month
  Muscle mass percentage will be calculated by using single-frequency BIA with eight-point tactile electrodes (Omron HBF-500 BIA, Omron Medizintechnik, Mannheim, Germany), whose reliability with DXA and MRI measurements was previously demonstrated will be used. This device uses an AC of 500 µA with a single frequency of 50 kHz and eight electrodes in a tetrapolar arrangement, requiring the subject to stand on metal footpads in bare feet and grasp a pair of electrodes fxed on a handle, with arms extended in front of the chest.
Visceral Fat Level | one month
  Visceral fat level will be calculated by using single-frequency BIA with eight-point tactile electrodes (Omron HBF-500 BIA, Omron Medizintechnik, Mannheim, Germany), whose reliability with DXA and MRI measurements was previously demonstrated will be used. This device uses an AC of 500 µA with a single frequency of 50 kHz and eight electrodes in a tetrapolar arrangement, requiring the subject to stand on metal footpads in bare feet and grasp a pair of electrodes fxed on a handle, with arms extended in front of the chest.

SECONDARY OUTCOMES:
Total daily EE (Kcal/day) | one month
  The Apple Watch 44 mm (5th generation) using watchOS 6 (Apple Inc., Cupertino, California, USA) will be used.
Hours/day spent upright | one month
  The Apple Watch 44 mm (5th generation) using watchOS 6 (Apple Inc., Cupertino, California, USA) will be used.
Number of strides and distance (Km) | one month
  The Apple Watch 44 mm (5th generation) using watchOS 6 (Apple Inc., Cupertino, California, USA) will be used.
Daily movement EE (Kcal/day) | one month
  The Apple Watch 44 mm (5th generation) using watchOS 6 (Apple Inc., Cupertino, California, USA) will be used to calculate.
EE (Kcal/min) | one month
  The Apple Watch 44 mm (5th generation) using watchOS 6 (Apple Inc., Cupertino, California, USA) will be used to calculate this outocome in four targeted conditions (typing, loading the dishwasher, sweeping and walking upstairs and downstairs).
sleep onset latency (minutes) | one month
  Actigraphy analysis will be performed for 1 week, using the wGT3X-BT device by ActiGraph (Pensacola, FL, USA). This device is a triaxial accelerometer measuring wrist acceleration in three orthogonal axes at a sampling frequency of 80 Hz. This device is waterproof, with a battery life of approximately 3 weeks. The device does not provide any feedback to the participants about their activity or sleep. The acceleration data collected by the device will be used to obtain the estimates of this outcome for the whole week.
total sleep time (minutes) | one month
  Actigraphy analysis will be performed for 1 week, using the wGT3X-BT device by ActiGraph (Pensacola, FL, USA). This device is a triaxial accelerometer measuring wrist acceleration in three orthogonal axes at a sampling frequency of 80 Hz. This device is waterproof, with a battery life of approximately 3 weeks. The device does not provide any feedback to the participants about their activity or sleep. The acceleration data collected by the device will be used to obtain the estimates of this outcome for the whole week.
wake time after sleep onset (minutes) | one month
  Actigraphy analysis will be performed for 1 week, using the wGT3X-BT device by ActiGraph (Pensacola, FL, USA). This device is a triaxial accelerometer measuring wrist acceleration in three orthogonal axes at a sampling frequency of 80 Hz. This device is waterproof, with a battery life of approximately 3 weeks. The device does not provide any feedback to the participants about their activity or sleep. The acceleration data collected by the device will be used to obtain the estimates of this outcome for the whole week.
sleep efficiency (percentage) | one month
  Actigraphy analysis will be performed for 1 week, using the wGT3X-BT device by ActiGraph (Pensacola, FL, USA). This device is a triaxial accelerometer measuring wrist acceleration in three orthogonal axes at a sampling frequency of 80 Hz. This device is waterproof, with a battery life of approximately 3 weeks. The device does not provide any feedback to the participants about their activity or sleep. The acceleration data collected by the device will be used to obtain the estimates of this outcome for the whole week.

CONTACTS AND LOCATIONS:
Locations (1):
- ITER Center for Balance and Rehabilitation Research, Guidonia, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Herdman SJ, Blatt PJ, Schubert MC. Vestibular rehabilitation of patients with vestibular hypofunction or with benign paroxysmal positional vertigo. Curr Opin Neurol. 2000 Feb;13(1):39-43. doi: 10.1097/00019052-200002000-00008. PMID 10719648
- [Background] Hall CD, Herdman SJ, Whitney SL, Anson ER, Carender WJ, Hoppes CW, Cass SP, Christy JB, Cohen HS, Fife TD, Furman JM, Shepard NT, Clendaniel RA, Dishman JD, Goebel JA, Meldrum D, Ryan C, Wallace RL, Woodward NJ. Vestibular Rehabilitation for Peripheral Vestibular Hypofunction: An Updated Clinical Practice Guideline From the Academy of Neurologic Physical Therapy of the American Physical Therapy Association. J Neurol Phys Ther. 2022 Apr 1;46(2):118-177. doi: 10.1097/NPT.0000000000000382. PMID 34864777
- [Background] Micarelli A, Viziano A, Pistillo R, Granito I, Micarelli B, Alessandrini M. Sleep Performance and Chronotype Behavior in Unilateral Vestibular Hypofunction. Laryngoscope. 2021 Oct;131(10):2341-2347. doi: 10.1002/lary.29719. Epub 2021 Jun 30. PMID 34191310
- [Background] Micarelli A, Viziano A, Micarelli B, Augimeri I, Alessandrini M. Vestibular rehabilitation in older adults with and without mild cognitive impairment: Effects of virtual reality using a head-mounted display. Arch Gerontol Geriatr. 2019 Jul-Aug;83:246-256. doi: 10.1016/j.archger.2019.05.008. Epub 2019 May 10. PMID 31102927
- [Background] Alessandrini M, Viziano A, Pistillo R, Granito I, Basso L, Preziosi N, Micarelli A. Changes in daily energy expenditure and movement behavior in unilateral vestibular hypofunction: Relationships with neuro-otological parameters. J Clin Neurosci. 2021 Sep;91:200-208. doi: 10.1016/j.jocn.2021.07.012. Epub 2021 Jul 17. PMID 34373028
- [Background] Micarelli A, Viziano A, Granito I, Micarelli RX, Felicioni A, Alessandrini M. Changes in body composition in unilateral vestibular hypofunction: relationships between bioelectrical impedance analysis and neuro-otological parameters. Eur Arch Otorhinolaryngol. 2021 Jul;278(7):2603-2611. doi: 10.1007/s00405-020-06561-z. Epub 2021 Jan 3. PMID 33392761
- [Background] Micarelli A, Viziano A, Augimeri I, Micarelli D, Alessandrini M. Three-dimensional head-mounted gaming task procedure maximizes effects of vestibular rehabilitation in unilateral vestibular hypofunction: a randomized controlled pilot trial. Int J Rehabil Res. 2017 Dec;40(4):325-332. doi: 10.1097/MRR.0000000000000244. PMID 28723718
- [Background] McKeown J, McGeoch PD, Grieve DJ. The influence of vestibular stimulation on metabolism and body composition. Diabet Med. 2020 Jan;37(1):20-28. doi: 10.1111/dme.14166. Epub 2019 Nov 8. PMID 31667892
- [Background] Fuller PM, Jones TA, Jones SM, Fuller CA. Neurovestibular modulation of circadian and homeostatic regulation: vestibulohypothalamic connection? Proc Natl Acad Sci U S A. 2002 Nov 26;99(24):15723-8. doi: 10.1073/pnas.242251499. Epub 2002 Nov 14. PMID 12434016
- [Background] McGeoch PD. Can Vestibular Stimulation be Used to Treat Obesity?: Vestibular stimulation targeting the otoliths could rebalance energy homeostasis to trigger a leaner body habitus and thus treat metabolic syndrome. Bioessays. 2019 Feb;41(2):e1800197. doi: 10.1002/bies.201800197. Epub 2019 Jan 7. PMID 30614540
- [Background] Fuller PM, Jones TA, Jones SM, Fuller CA. Evidence for macular gravity receptor modulation of hypothalamic, limbic and autonomic nuclei. Neuroscience. 2004;129(2):461-71. doi: 10.1016/j.neuroscience.2004.05.059. PMID 15501603
- [Background] Tighilet B, Chabbert C. Adult neurogenesis promotes balance recovery after vestibular loss. Prog Neurobiol. 2019 Mar;174:28-35. doi: 10.1016/j.pneurobio.2019.01.001. Epub 2019 Jan 15. PMID 30658127